CLINICAL TRIAL: NCT02869867
Title: Does the Application of Cold Decreases the Pain Associated in the Pose of a Patch of Capsaicine at High Concentration on the Carrier Patients of Localized Neuropathic Pains ? - DIDOCAP
Acronym: DIDOCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHD049-16
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Results first posted 2024-08-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Localized Neuropathic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qutenza® without refrigerated cushion (No Intervention): Qutenza® without refrigerated cushion
- Qutenza® with refrigerated cushion (Experimental): Qutenza® with refrigerated cushion
  Interventions: Other: refrigerated cushion

INTERVENTIONS:
Other: refrigerated cushion — refrigerated cushion
  Arms: Qutenza® with refrigerated cushion

SUMMARY:
Nursing study, prospective, randomized, two-center open-label.

Patients will be randomized into two groups during their first laying Qutenza®:

* Patients receiving the laying of Qutenza® without refrigerated cushion
* Patients receiving the laying of Qutenza® associated with a refrigerated cushion

The objective of the study is to evaluate the effectiveness of the application of cold to the reduction of pain (burning) after one hour of patch installation high concentration capsaicin (Qutenza®) in patients localized neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Major
* Do not opposing the participation in the study
* Monitoring in the case of localized neuropathic pain
* Diagnostic with neuropathic pain score ≥ 4
* Neuropathic pain conventional treatment failure of first-line
* Front advantage of laying a first patch Qutenza®
* With ability to understand the proposed study

Exclusion Criteria:

* Patch Installation on the feet, face, mucous membranes
* Eutectic mixture of local anesthetics (EMLA) Pose premedication
* Having Already received prior to the installation of a patch of Qutenza®
* Allergy to components Qutenza®
* Known and poorly stabilized hypertension
* Known cryoglobulinaemia
* Pregnant or lactating women
* Patient enjoying a measure of legal protection (guardianship, guardianship ...)
* Private Patient freedom
* No affiliation to a social security scheme.
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHLVO de Challans, Challans
  - CHD Vendée de la Roche sur Yon, La Roche-sur-Yon
  - Clinique Brétéché, Nantes

REFERENCES:
- [Result] Tailliez N, Planche L, Dorion A, Kacki N, Dimet J, Pluchon YM. Effect of Cooling Capsaicin Application Site on Reducing Burning Sensation in Neuropathic Pain Patients: A Randomized Controlled Trial. Pain Manag Nurs. 2025 Apr;26(2):e159-e164. doi: 10.1016/j.pmn.2024.09.001. Epub 2024 Nov 12. PMID 39532578

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Qutenza® without refrigerated cushion | Qutenza® with refrigerated cushion
Started | 50 | 50
Completed | 44 | 45
Not Completed | 6 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Population: All analyses were performed according to the intention-to-treat principle by including all randomized patients to whom the Qutenza® patch was applied.
Groups:
- Total: Total of all reporting groups
Arm/Group | Qutenza® Without Refrigerated Cushion | Qutenza® With Refrigerated Cushion | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12) | 49 (14) | 50 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 40 | 74
  Male | 15 | 10 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Pain Scale (Burning Pain)
Description: Burning pain will be estimated by the patient using a non-graduated 10 cm line, presented horizontally to the patient with the extreme position of the vertical border on the left (0mm) representing the absence of perceived pain and the extreme position on the right (10 cm), the perception of the maximum pain that the patient can imagine. The information obtained is measured and translated into a score between 0 and 10.
  The patient will be asked: "How would you rate the intensity of pain caused by Qutenza patch application?
Time Frame: after 1 hour of installation of Qutenza patch
Population: Intent to treat Population (all participants who received a Qutenza patch)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Qutenza® without refrigerated cushion | Qutenza® with refrigerated cushion
Number analyzed (Participants) | 49 | 50
units on a scale | 6.99 [6.2 to 7.77] | 3.78 [3 to 4.56]
Statistical Analysis 1: Comparison: Qutenza® without refrigerated cushion vs Qutenza® with refrigerated cushion; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 3.20, 95% CI 2-sided [2.09 to 4.31]

ADVERSE EVENTS:
Description: Death, serious adverse events and other (non serious adverse events) were not assessed for the study
Arm/Group | Qutenza® without refrigerated cushion | Qutenza® with refrigerated cushion
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT02869867/Prot_SAP_000.pdf